CLINICAL TRIAL: NCT04666610
Title: A Randomized, Dose-Finding and Confirmatory, Double-Blind, Placebo-Controlled, Parallel-Group Multicenter Study With a 2 Stage Adaptive Design and Randomized Withdrawal to Evaluate the Efficacy, Safety, and Tolerability of Brivaracetam as Monotherapy in Patients 2 to 25 Years of Age With Childhood Absence Epilepsy or Juvenile Absence Epilepsy
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of Brivaracetam as Monotherapy in Patients 2 to 25 Years of Age With Childhood Absence Epilepsy or Juvenile Absence Epilepsy
Acronym: EXPAND
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01269; 2020-002750-24 (EudraCT Number); 2023-510428-55-00 (Registry Identifier: CTIS); U1111-1303-2521 (Other: Universal Trial Number (UTN))
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Childhood Absence Epilepsy; Juvenile Absence Epilepsy
Keywords: Brivaracetam; Briviact; Epilepsy; Childhood absence Epilepsy; Juvenile absence epilepsy; CAE; JAE
MeSH Terms: conditions — Epilepsy, Absence; Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Brivaracetam 200 mg (Experimental): Placebo-Controlled (PC) and Active Treatment (AT) Period:
  Stage 1: Study participants randomized to brivaracetam (BRV) 200mg/day (or equivalent dose) will receive these doses during the 2-week PC period and subsequent 11-week AT period.
  Interventions: Drug: Brivaracetam
- Placebo to 200 mg brivaracetam (Experimental): Placebo-Controlled (PC) and Active Treatment (AT) Period:
  Stage 1: Study participants randomized to 'placebo to BRV 200mg/day' (or equivalent dose) will receive placebo during the PC period followed by BRV 200mg/day (or equivalent dose) during the AT period.
  Interventions: Drug: Brivaracetam; Other: Placebo
- Brivaracetam 100 mg (Experimental): Placebo-Controlled (PC) and Active Treatment (AT) Period:
  Stage 1: Study participants randomized to BRV 100mg/day (or equivalent dose) will receive these doses during the 2-week PC period and subsequent 11-week AT period.
  Interventions: Drug: Brivaracetam
- Placebo to 100 mg brivaracetam (Experimental): Placebo-Controlled (PC) and Active Treatment (AT) Period:
  Stage 1: Study participants randomized to 'placebo to BRV 100mg/day' (or equivalent dose) will receive placebo during the PC period followed by BRV 100mg/day (or equivalent dose) during the AT period.
  Interventions: Drug: Brivaracetam; Other: Placebo
- Optimal dose of BRV (defined following Stage 1) (Experimental): Placebo-Controlled (PC) and Active Treatment Period (AT):
  Stage 2: Study participants will be randomized in Stage 2 to receive a fixed dose of the optimal dose of brivaracetam (defined following Stage 1). Study participants randomized to the BRV optimal dose will receive this dose during the 2-week PC period and subsequent 11-week AT period.
  Interventions: Drug: Brivaracetam
- Placebo to BRV optimal dose (defined following Stage 1) (Experimental): Placebo-Controlled (PC) and Active Treatment (AT) Period:
  Stage 2: Study participants will be randomized in Stage 2 of the study to 'placebo to BRV optimal dose'. Study participants randomized to placebo to brivaracetam (BRV) optimal dose will receive placebo during the PC period followed by BRV optimal dose during the AT period.
  Interventions: Drug: Brivaracetam; Other: Placebo
- Brivaracetam received during RDW (Experimental): Randomized Withdrawal (RDW) Period:
  Only study participants who are absence seizure-free based on the outcome of the 24h EEG of Visit 5 will enter the RDW Period. Participants who are randomized to this arm will continue on the Brivaracetam dose they were receiving in the AT period.
  Interventions: Drug: Brivaracetam
- Placebo received during RDW (Experimental): Randomized Withdrawal (RDW) Period:
  Only study participants who are absence seizure-free based on the outcome of the 24h EEG of Visit 5 will enter the RDW Period. Study participants who are randomized to the placebo arm in the RDW Period will be tapered down to 0 mg and receive 0 mg for 2 weeks.
  Interventions: Drug: Brivaracetam; Other: Placebo

INTERVENTIONS:
Drug: Brivaracetam — * Pharmaceutical form: Oral solution
  * Route of administration: Oral use
  Brivaracetam (oral solution [10 mg/ml, 5 mg/ml or 2.5 mg/ml] will be administered.
  Other Names: BRV
Other: Placebo — Subjects will receive placebo at pre-specified time-points to maintain the blinding.
  Other Names: PBO
  Arms: Placebo received during RDW; Placebo to 100 mg brivaracetam; Placebo to 200 mg brivaracetam; Placebo to BRV optimal dose (defined following Stage 1)

SUMMARY:
The purpose of the study is to test the efficacy, safety and tolerability of brivaracetam monotherapy in study participants 2 to 25 years of age inclusive with childhood absence epilepsy (CAE) or juvenile absence epilepsy (JAE).

ELIGIBILITY:
Inclusion Criteria:

* Study participant is 2 to 25 years of age inclusive, at the time of signing the informed consent. No study participants from 2 to <4 years of age will be included in Stage 1
* Study participant is diagnosed with either childhood absence epilepsy (CAE) or juvenile absence epilepsy (JAE) as defined by the International League Against Epilepsy (ILAE) criteria
* Study participants 2 to <4 years of age and participants who had onset of absence seizures at an age younger than 4 years must have a negative glucose transporter type 1 deficiency syndrome (GLUT1DS) genetic test
* Study participant is untreated with antiepileptic drugs (AEDs) or pretreated for absence seizures with a maximum of 2 historical AEDs, but without AED treatment for a period of at least 5 half-lives of the AED before randomization into this study. The UCB study physician should be consulted if in doubt
* Study participant has electroencephalogram (EEG) evidence of bilateral synchronous, symmetric generalized paroxysmal spike waves (2.5-6 hertz) with normal background activity and with at least 1 electrographically recorded seizure lasting 3 seconds or more on a 1-hour EEG with hyperventilation (HV) while awake at Visit 1 (V1), or on a historical EEG up to 12 weeks before enrollment
* Study participant has a history of clinically evident absence seizures occurring on at least 3 days per week in the 2 weeks prior to enrollment
* Study participant is without treatment with psychoactive drugs or on a stable dose for at least 2 weeks prior to randomization
* Study participant has normal neurological examination, head size, development and cognition
* Body weight is ≥9 kg
* Male and female

  a) A sexually active male study participant must agree to use contraception during the treatment period and for at least 2 days, corresponding to the time needed to eliminate study treatment, after the last dose of study treatment and refrain from donating sperm during this period b) A female study participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies: The study participant is premenarchial OR A woman of childbearing potential (WOCBP) who agrees to follow the contraceptive guidance during the treatment period and for at least 2 days after the last dose of study treatment, corresponding to the time needed to eliminate study treatment
* Study participant provides consent/assent, and the study participant's parent/legal representative/caregiver provides signed informed consent for minor study participants, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

* Study participant has a history of nonfebrile seizures other than absence seizures (eg, generalized tonic-clonic seizures or myoclonic seizures)
* Study participant has a history of absence status epilepticus
* Study participant has a history or presence of paroxysmal nonepileptic seizures
* Study participant has a clinically relevant electrocardiogram (ECG) abnormality in the opinion of the Principal Investigator
* Study participant has hepatic impairment (Child Pugh Score A, B, or C) based on the Investigator's assessment
* Study participant has a history of major psychiatric disease or any clinically significant medical condition that would preclude appropriate study participation
* Study participant has active suicidal ideation prior to study entry as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS; for study participants 6 years or older) or clinical judgement (for study participants younger than 6 years). The study participant should be referred immediately to a Mental Healthcare Professional
* Study participant has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt). The study participant should be immediately evaluated by a Mental Healthcare Professional to address safety concerns
* Study participant with known fructose intolerance or hypersensitivity of any of the ingredients in brivaracetam oral solution
* Study participant has end-stage kidney disease requiring dialysis
* Concomitant use of rifampicin/rifampin; prior use must have been stopped at least 2 months before randomization
* Concomitant use of strong CYP2C19 inhibitors like fluconazole, fluoxetine and fluvoxamine, prior use must have been stopped at least 1 week before randomization
* Study participant has participated in another study of an investigational medicinal product (IMP; and/or an investigational device) within the previous 30 days prior to informed consent
* Study participant has clinical or EEG findings not consistent with a diagnosis of childhood absence epilepsy (CAE) or juvenile absence epilepsy (JAE)

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who met the criteria for absence seizure freedom within 4 days prior to or during the 24-hour ambulatory electroencephalogram (EEG) at Day 14 | Day 14
  A 24-hour ambulatory electroencephalogram (EEG) will be performed at day 14. The awake hours from the EEG will be analyzed for absence seizures. Every 24-hour EEG will include hyperventilation as a standard provocation test at the beginning of the EEG. Patient will be regarded as not meeting the criteria for absence seizure freedom if they received benzodiazepine in the 4 days prior to the EEG or during the EEG.

SECONDARY OUTCOMES:
Percentage of participants who met the criteria for absence seizure freedom during the randomized withdrawal (RDW) period as determined by electroencephalogram (EEG) | From Week 13 to Week 17
  Study participants (or their care givers) who believe they are experiencing a recurrence of absence seizures will contact the clinical site for a 1-hour EEG (with hyperventilation (HV)). If no absence seizure is observed during this 1hr EEG (locally read), the study participant will receive a 24-hour ambulatory EEG. If an absence seizure is observed during either EEG, the study participant will be considered as not Absence seizure free and leave the study. If no absence seizures are determined by 1/24hr ambulatory EEG the participant will conduct a 24-hour EEG at week 17. Patient will be regarded as not meeting the criteria for absence seizure freedom if they received benzodiazepine in the 4 days prior to the EEG or during the EEG.
  The awake hours from the EEG will be analyzed for absence seizures. Every 24-hour EEG will include HV as a standard provocation test at the beginning of the EEG.
Percent change from Baseline to Day 14 in number of absence seizures on 24-hour ambulatory electroencephalogram (EEG) | From Baseline to Day 14
  A 24-hour ambulatory electroencephalogram (EEG) will be performed at baseline and day 14. The awake hours from the EEG will be analyzed for absence seizures. Every 24-hour EEG will include hyperventilation as a standard provocation test at the beginning of the EEG.
  This endpoint is the difference between the number of seizures at baseline and Day 14.
Percentage of participants who met the criteria for absence seizure freedom based on diary during the 4 days prior to the visit at Day 14 | Day 14
  During the study subjects will keep a diary to record daily seizure activity from Visit 1 until end of the randomized withdrawal (RDW) Period. Each seizure type experienced will be recorded. The last 4 study days prior to Day 14 EEG are used for this endpoint.
  Patient will be regarded as not meeting the criteria for absence seizure freedom if they received benzodiazepine in the 4 days prior to the EEG or during the EEG.
Percentage of participants who met the criteria for absence seizure freedom on 24-hour ambulatory electroencephalogram (EEG) at Week 12 | Week 12
  A 24-hour ambulatory electroencephalogram (EEG) will be performed at day 14. The awake hours from the EEG will be analyzed for absence seizures. Every 24-hour EEG will include hyperventilation as a standard provocation test at the beginning of the EEG. Patient will be regarded as not meeting the criteria for absence seizure freedom if they received benzodiazepine in the 4 days prior to the EEG or during the EEG.
Percentage of participants who met the criteria for absence seizure freedom based on diary during the 4 days prior to the visit at Week 12 | Week 12
  During the study subjects will keep a diary to record daily seizure activity from Visit 1 until end of the randomized withdrawal (RDW) Period. Each seizure type experienced will be recorded. The last 4 study days prior to Week 12 EEG are used for this endpoint. Patient will be regarded as not meeting the criteria for absence seizure freedom if they received benzodiazepine in the 4 days prior to the EEG or during the EEG.
Percentage of participants with treatment-emergent adverse events (TEAEs) during the study | From Day 1 until End of Safety Follow-Up (up to Week 23)
  An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medicinal product (IMP).
Percentage of participants with treatment-emergent adverse events (TEAEs) leading to discontinuation of study treatment | From Day 1 until End of Down Titration Period (up to Week 21)
  An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medicinal product (IMP).
Percentage of participants with serious adverse events (SAEs) during the study | From Screening Period (Day -14 to Day -2) until End of Safety Follow-Up (up to Week 23)
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Results in permanent or significant disability/incapacity
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
Percentage of participants with drug-related treatment-emergent adverse events (TEAEs) during the study | From Baseline (Day -1) until End of Safety Follow-Up (up to Week 23)
  An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medicinal product (IMP). 'Drug related AEs' are the subset of AEs that the investigator considers as related to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (53):
- United States (12):
  - N01269 115, Birmingham, Alabama
  - N01269 118, Long Beach, California
  - N01269 105, Orange, California
  - N01269 116, Denver, Colorado
  - N01269 103, Loxahatchee Groves, Florida
  - N01269 111, Miami, Florida
  - N01269 101, Tampa, Florida
  - N01269 104, Winter Park, Florida
  - N01269 110, Augusta, Georgia
  - N01269 100, New Brunswick, New Jersey
  - N01269 109, Winston-Salem, North Carolina
  - N01269 106, Philadelphia, Pennsylvania
- Australia (4):
  - N01269 203, Heidelberg
  - N01269 202, Melbourne
  - N01269 200, Randwick
  - N01269 201, South Brisbane
- Belgium (2):
  - N01269 301, Brussels
  - N01269 300, Edegem
- Georgia (5):
  - N01269 400, Tbilisi
  - N01269 401, Tbilisi
  - N01269 402, Tbilisi
  - N01269 403, Tbilisi
  - N01269 405, Tbilisi
- Italy (7):
  - N01269 323, Messina
  - N01269 321, Milan
  - N01269 324, Milan
  - N01269 320, Pavia
  - N01269 322, Roma
  - N01269 325, Roma
  - N01269 326, Verona
- Poland (5):
  - N01269 533, Gdansk
  - N01269 530, Krakow
  - N01269 534, Lodz
  - N01269 531, Lublin
  - N01269 532, Warsaw
- Romania (4):
  - N01269 562, Bucharest
  - N01269 563, Bucharest
  - N01269 560, Iași
  - N01269 561, Timişoara, Judeţ Timiş
- Slovakia (3):
  - N01269 632, Bardejov
  - N01269 630, Dubnica nad Váhom
  - N01269 631, Nové Zámky
- Spain (3):
  - N01269 351, Madrid
  - N01269 353, Seville
  - N01269 354, Terrassa
- Ukraine (8):
  - N01269 600, Dnipro
  - N01269 601, Dnipro
  - N01269 604, Kharkiv
  - N01269 608, Kharkiv
  - N01269 603, Kyiv
  - N01269 606, Kyiv
  - N01269 607, Uzhhorod
  - N01269 602, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Bast T, Schulz AL, Floricel F, Morita D, Cleveland JM, Elshoff JP. Efficacy and tolerability of brivaracetam monotherapy in childhood and juvenile absence epilepsy: An innovative adaptive trial design. Epilepsia Open. 2022 Dec;7(4):588-597. doi: 10.1002/epi4.12628. Epub 2022 Aug 4. PMID 35844134